CLINICAL TRIAL: NCT07176221
Title: Safety and Efficacy of Endoscopic Cardial Constriction Ligation （ECCL） With a Novel Disposable Endoscope: A Multicenter Randomized Controlled Trial
Brief Title: Endoscopic Cardial Constriction Ligation (ECCL) for Refractory GERD Using a Disposable Endoscope
Acronym: ECCL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ying Zhu (Other)
Responsible Party: Sponsor-Investigator, Ying Zhu, Principal Investigator, Clinical Professor, Shenzhen Hospital of Southern Medical University
Organization: Shenzhen Hospital of Southern Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NYSZYYEC2025K055R002
Record Dates: First submitted 2025-08-16; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal Reflux Disease (GERD).; Endoscopic cardia constriction ligation (ECCL); novel disposable endoscope
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will undergo endoscopic cardia constriction ligation (ECCL) using disposable endoscopes. The procedure involves: under direct visualization, sequentially suctioning and ligating one ring each on the lesser curvature, posterior wall, and greater curvature of the cardia, capturing the mucosal and muscular layers. A hemostatic clip will be used to secure the base of the ligated tissue on the greater curvature. Six hours post-procedure, patients may consume lukewarm liquid or semi-liquid diets and continue acid-suppressive therapy for two weeks. Vital signs and any procedure-related serious adverse events will be recorded for statistical analysis.
  Interventions: Procedure: endoscopic cardia constriction ligation
- Control Group (Active Comparator): The control group will undergo endoscopic cardia constriction ligation (ECCL) using traditional endoscopes. The procedure involves: under direct visualization, sequentially suctioning and ligating one ring each on the lesser curvature, posterior wall, and greater curvature of the cardia, capturing the mucosal and muscular layers. A hemostatic clip will be used to secure the base of the ligated tissue on the greater curvature. Six hours post-procedure, patients may consume lukewarm liquid or semi-liquid diets and continue acid-suppressive therapy for two weeks. Vital signs and any procedure-related serious adverse events will be recorded for statistical analysis.
  Interventions: Procedure: endoscopic cardia constriction ligation

INTERVENTIONS:
Procedure: endoscopic cardia constriction ligation — The experimental group used disposable endoscopes to perform ECCL, while the control group used traditional endoscopes to perform ECCL. ECCL involves ligating and fixing the mucosa and partial muscle layer above the dentate line under direct endoscopic visualization to create folds. Post-procedure, the ligated mucosa undergoes ischemic necrosis and heals to form scar tissue, thereby reducing the cardia diameter, increasing LES pressure, and alleviating reflux symptoms.

SUMMARY:
This study will recruit patients aged 18-80 with refractory gastroesophageal reflux disease (GERD). These patients had a disease course of more than six months, experienced typical symptoms such as acid reflux and heartburn, and had no symptom relief after taking a double dose of acid-suppressing medication for eight consecutive weeks. All eligible participants will undergo Endoscopic Cardial Constriction Ligation (ECCL) using a disposable endoscope. The procedure will follow a standardized protocol: mucosal and muscle layers of the cardia will be ligated at the lesser curvature, posterior wall, and greater curvature, with the ligated tissue at the greater curvature secured by a hemostatic clip. All patients will receive acid-suppressing therapy post-surgery and will be followed up at three and six months. The follow-ups will assess their GERD-Q scores, symptom relief, and incidence of complications.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a common digestive disorder, with endoscopic manifestations including non-erosive reflux disease (NERD), reflux esophagitis (RE), and Barrett's esophagus (BE). Typical symptoms include heartburn and regurgitation, while atypical symptoms encompass chest pain, epigastric pain, belching, and extraesophageal symptoms. Epidemiological surveys in China indicate a prevalence of heartburn occurring at least once weekly ranging from 1.9% to 7.0%. Chronic, recurrent GERD significantly impairs patients' quality of life and may increase the risk of Barrett's esophagus, esophageal mucosal dysplasia, and esophageal adenocarcinoma. The etiology of GERD is complex, involving increased esophageal acid exposure, lower esophageal sphincter (LES) relaxation, low esophagogastric junction (EGJ) pressure, impaired esophageal clearance, hiatal hernia, and damage to the mucosal barrier by cytokines (e.g., IL-6, IL-8, platelet-activating factor PAF) and other factors.

Currently, the first-line treatment for GERD includes lifestyle modifications and oral acid-suppressive medications, such as proton pump inhibitors (PPIs) and potassium-competitive acid blockers (P-CABs). However, some patients with refractory GERD require long-term acid-suppressive therapy, and prolonged PPI use may increase the risk of Clostridioides difficile infection, community-acquired pneumonia, gastric cancer, and chronic kidney disease, while short-term P-CAB use may lead to hypergastrinemia [13]. According to the 2020 Chinese GERD Expert Consensus, for patients with refractory GERD who fail medical therapy, endoscopic or surgical treatment may be considered after excluding other causes and confirming evidence of reflux.

Traditional endoscopes are reusable and require cleaning and disinfection after each use, but complete sterilization may not always be achieved, posing a risk of cross-infection. In contrast, disposable endoscopes eliminate the risk of cross-infection, bypass the need for cleaning and disinfection, and reduce the incidence of instrument-related infections, while offering comparable functionality and operability to traditional endoscopes. Endoscopic cardia constriction ligation (ECCL) is an emerging endoscopic treatment technique, first performed by Professor Linghu Enqiang in 2013. This procedure involves ligating and fixing the mucosa and partial muscle layer above the dentate line under direct endoscopic visualization, creating mucosal folds. Post-procedure, the ligated mucosa undergoes ischemic necrosis and heals to form scar tissue, reducing the cardia diameter, increasing LES pressure, and alleviating reflux symptoms. ECCL is characterized by simple operation and minimal invasiveness, making it safer than traditional surgical procedures. Related complications, such as bleeding after ligation band detachment and retrosternal pain, are infrequent, resolve quickly, and no severe adverse events have been reported to date. However, the long-term efficacy of ECCL requires further validation.

Currently, there are no studies on the efficacy and safety of ECCL performed using disposable endoscopes. This study aims to conduct a randomized controlled trial to compare the effectiveness, safety, flexibility, and imaging clarity of ECCL performed with disposable versus traditional endoscopes in treating refractory GERD, providing scientific evidence to optimize treatment strategies and inform future GERD treatment guidelines.

Participants in this study will be randomly assigned to either the disposable endoscope group or the traditional endoscope group to undergo ECCL treatment. The primary objective is to compare the efficacy of ECCL performed with disposable versus traditional endoscopes in treating refractory GERD. Secondary objectives include: 1) Evaluating the observation clarity, flexibility, and compatibility of disposable endoscopes with surgical consumables; 2) Assessing the incidence of device failures and complications related to disposable endoscope-guided ECCL, such as mucosal injury, bleeding, and perforation.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 18-80 years;
* (2) Disease duration ≥6 months, with typical symptoms such as acid regurgitation and heartburn, and a confirmed diagnosis of GERD;
* (3) GERD patients whose symptoms are not relieved after 8 weeks of continuous double-dose acid-suppressive therapy;
* (4) Willing to participate in the study and have signed the informed consent form.

Exclusion Criteria:

* (1) Patients with precancerous lesions such as early esophageal cancer or Barrett's esophagus >3 cm, or advanced upper gastrointestinal cancer identified on endoscopy;
* (2) Patients with hiatal hernia ≥2 cm, severe reflux esophagitis (LA-C or LA-D grade), esophageal or gastric varices, esophageal ulcer or stenosis, or a history of esophageal or gastric surgery;
* (3) Patients with esophageal motility disorders such as achalasia or diffuse esophageal spasm, rheumatic diseases such as systemic sclerosis or Sjögren's syndrome, or eosinophilic esophagitis;
* (4) Patients with a history of endoscopic or surgical anti-reflux procedures;
* (5) Patients with coagulation disorders, severe cardiopulmonary diseases, or inability to tolerate anesthesia, endoscopy, or treatment;
* (6) Women in the puerperium.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in GERD-Q Score | From baseline before the procedure to 6 months post-procedure
  Change in GERD-Q score (a validated questionnaire assessing GERD-related symptoms such as acid regurgitation and heartburn) from baseline, measured in patients undergoing ECCL with disposable endoscopes versus traditional endoscopes. GERD-Q scores are collected at baseline (pre-procedure via questionnaire and endoscopic examination), 3 months post-procedure, and 6 months post-procedure during follow-up visits.

SECONDARY OUTCOMES:
Rate of Clinical Feasibility of ECCL Treatment Using Disposable Endoscopes | From baseline before the procedure to 6 months post-procedure
  After passing through the cardia, the endoscope can be successfully inverted to observe the cardia, clearly visualizing the dentate line. During endoscopic cardia constriction ligation (ECCL), the ligation device can be securely attached to the endoscope, effectively suctioning the gastric wall mucosa and smoothly releasing the ligation ring. Additionally, all abnormal findings mentioned in the gastroscopy report should be photographed and documented.
  If the entire gastroscopy examination and treatment are completed, it is considered feasible.
  If the examination or treatment is interrupted due to issues with the endoscope itself, it is considered infeasible.
  Calculation Formula: Clinical feasibility rate = (Number of participants completing the procedure successfully ÷ Total number of participants) × 100%Clinical feasibility rate of disposable endoscope ECCL treatment = (Number of participants completing the procedure successfully ÷ Total number of participants) × 100%.
Device Failure/Defect Rate | From baseline before the procedure to 6 months post-procedure
  Observe whether the device experiences any malfunctions during the procedure, such as image interruption, blockage, or leakage during water delivery.
Number of Participants with Endoscope-Related Mucosal Injury | From baseline before the procedure to 1 hour post-procedure
  Document any occurrences of mucosal injury directly related to the use of disposable endoscopes during the ECCL procedure.
Number of Participants with Gastrointestinal Perforation | From baseline before the procedure to 1 hour post-procedure
  Record any cases of gastrointestinal perforation occurring during or within 1 hour after the ECCL procedure using disposable endoscopes.
Number of Participants with Significant Bleeding | From baseline before the procedure to 1 hour post-procedure
  Identify participants who experience significant bleeding during or within 1 hour post-procedure.
Number of Participants with Procedure-Related Adverse Reactions | From baseline before the procedure to 6 months post-procedure
  Track adverse reactions such as pain, bleeding, or infection occurring after the ECCL procedure.
Number of Participants With Clear Endoscopic Image Quality During ECCL Procedure | Time Frame: From baseline before the procedure to end of procedure
  Image clarity will be assessed based on the ability to accurately identify the dentate line of the cardia.
  Grade A: Brightness, contrast, and sharpness are sufficient to clearly identify the dentate line.
  Grade B: Poor brightness, contrast, or sharpness prevents identification of the dentate line. Participants graded as "A" will be counted. Unit of Measure: Number of Participants
Number of Participants With Satisfactory Endoscope Flexibility During ECCL Procedure | Time Frame: From baseline before the procedure to end of procedure
  Flexibility will be assessed based on the ability to perform retroflexion smoothly.
  Grade A: Endoscope can be retroflexed smoothly.
  Grade B: Endoscope cannot be retroflexed smoothly. Participants graded as "A" will be counted. Unit of Measure: Number of Participants
Number of Participants With Compatible Consumables During ECCL Procedure | From baseline before the procedure to end of procedure
  Compatibility will be assessed based on successful attachment and operation of ligation devices.
  Grade A: Endoscope is compatible with ligation device; procedure proceeds smoothly.
  Grade B: Endoscope is incompatible with ligation device; procedure cannot proceed. Participants graded as "A" will be counted. Unit of Measure: Number of Participants
Composite Success Rate of ECCL Using Disposable Endoscopes | From baseline before the procedure to 6 months post-procedure
  Composite success is defined as a case in which all three procedural parameters are graded as "A":
  Image clarity sufficient to identify the dentate line of the cardia
  Endoscope flexibility allowing smooth retroflexion
  Compatibility of the endoscope with ligation devices enabling uninterrupted operation
  If any parameter is graded "B", the case is considered unsuccessful. Success rate is calculated as: (Number of Successful Cases / Total Number of Participants in Group) × 100 Unit of Measure: Percentage of Participants

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT07176221/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT07176221/ICF_001.pdf